CLINICAL TRIAL: NCT02234700
Title: To Estimate Whether Corneal Epithelial Defects Occur in Patients With Acquired Nasolacrimal Duct Obstructions is Linked to Changes Occurring Within Ocular Bacterial Flora in These Patients, and What Are the Specific Changes in Their Flora.
Brief Title: Are Corneal Epithelial Defects Related to Changes in Ocular Bacterial Flora in Patients With ANLDO
Acronym: ANLDO
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Sponsor
Other Study IDs: TASMC-14-AA-0071-CTIL
Record Dates: First submitted 2014-08-26; First posted 2014-09-09 (Estimated); Last update posted 2014-09-09 (Estimated); Status verified 2014-09

CONDITIONS: Acquired Nasolacrimal Duct Obstruction

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: None Retained — Bacterial flora from the eye
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Comparison between patients with nasolacrimal duct obstruction and healthy patients and the influence of their bacterial flora on the corneal epithelium.

DETAILED DESCRIPTION:
Any patient with nasolacrimal duct obstruction above the age of 18 Comparing changes in their bacterial ocular flora to healthy patients without obstruction and above 18 years of age

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, nasolacrimal duct obstruction

Exclusion Criteria:

* younger then 18 years of age
* ocular infections
* patients after repair of lacrimal duct surgery
* systemic active diseases
* patients taking medication that are know to influence bacterial flora of the eye

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 30 patients with nasolacrimal duct obstruction and 30 healthy patients
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2014-08; Primary Completion 2015-02 (Estimated); Study Completion 2015-02 (Estimated)

PRIMARY OUTCOMES:
the change of ocular normal flora in patients with nasolacrimal duct obstruction as a comparison to general population. | 6 month
  as the literature suggests most of the ocular flora is composed of Staphylococcus and Haemophilus, any change in these composition will be considered abnormal.

CONTACTS AND LOCATIONS:
Overall Officials: Yanir Kassif, M.D, Study Chair — Medical Center of the Galilee
Locations (1):
- Western Galileeh Hospital, Naharya, Israel